CLINICAL TRIAL: NCT00006003
Title: A Phase II Trial of SU5416 (NSC #696819) in Patients With Metastatic Melanoma
Brief Title: SU5416 in Treating Patients With Metastatic Melanoma That Has Been Previously Treated
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02346; 10395; N01CM17102 (NIH); CDR0000068011 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Semaxinib

ARMS (1):
- Treatment (semaxanib) (Experimental): Patients receive SU5416 IV over 60 minutes twice weekly for 4 weeks. Treatment continues for a minimum of 2 courses in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: semaxanib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: semaxanib — Given IV
  Other Names: semoxind; SU5416; Sugen 5416
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
SU5416 may stop the growth of malignant melanoma by stopping blood flow to the tumor. Phase II trial to study the effectiveness of SU5416 in treating patients who have metastatic melanoma that has been previously treated

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective response rate and stabilization of disease rates of patients with previously treated metastatic melanoma treated with SU5416.

II. Determine the toxicity of SU5416 in this patient population. III. Determine the median and overall survival and time to progression in these patients receiving this treatment.

OUTLINE: This is a multicenter study.

Patients receive SU5416 IV over 60 minutes twice weekly for 4 weeks. Treatment continues for a minimum of 2 courses in the absence of unacceptable toxicity or disease progression.

Patients are followed weekly for 4 weeks.

PROJECTED ACCRUAL: A total of 14-35 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed melanoma with documented metastatic disease

  * In transit metastases allowed
  * Lesion accessible for biopsy
* Measurable disease

  * Greater than 20 mm by conventional techniques ORgreater than 10 mm by spiral CT
* Documented progressive disease by radiologic study or physical examination
* Known history of CNS metastasis who have had treatment, are neurologicallystable, and do not require intravenous antibiotics or anticonvulsants eligibleprovided oral steroids are not required and brain scan (CT or MRI) showsabsence of active or residual disease

  * If neurologic signs or symptoms suggestive of CNS metastasis, negative brain scan required
* Performance status - WHO 0-2
* At least 12 weeks
* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 mg/dL
* Transaminases no greater than 2.5 times upper limit of normal
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* No uncompensated coronary artery disease
* No history of myocardial infarction or severe/unstable angina within past 6 months
* No severe peripheral vascular disease associated with diabetes mellitus
* No deep venous or arterial thrombosis within past 3 months
* No pulmonary embolism within past 3 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other significant uncontrolled underlying medical or psychiatric illness
* No serious active infections
* No other malignancy within past 5 years except for curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix
* No history of severe allergic or anaphylactic reactions to paclitaxel or docetaxel
* No other concurrent chemotherapy
* No other concurrent investigational antineoplastic drugs
* See Disease Characteristics
* No prior radiotherapy to only site of measurable disease
* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy
* No greater than 1 prior therapy for metastatic disease
* At least 4 weeks since prior therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2000-07; Primary Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Complete response rate | Up to 3 years
Overall response rate (complete and partial responses) | Up to 3 years
Maintenance of stable disease | Up to 3 years
Treatment toxicity | Up to 4 weeks post treatment
Time to progression | Up to 3 years
  Kaplan-Meier estimates will be calculated.
Survival | Up to 3 years
  Kaplan-Meier estimates will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gajewski, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States